CLINICAL TRIAL: NCT01822873
Title: Evaluation of Visual Function Impairments in Patients With Early Dry Age-related Macular Degeneration
Brief Title: Study on Visual Function Impairments in Dry Age-related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00036248
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-02

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal
- Age-related macular degeneration

SUMMARY:
The study hypothesis is that patients with dry age-related macular degeneration experience visual function impairments such as defects in dark adaptation, glare intolerance, poor light transition and reading in low lighting conditions. Studies have shown that patients in the early phases of AMD with normal visual acuity commonly reported difficulty with these visual functions but there have been no systematic studies evaluating these deficits in this population.

This prospective, exploratory study will include up to 130 patients with dry AMD and 60 controls. These patients will undergo the following non-invasive visual function testing:

* microperimetry with eye tracking
* low luminance visual acuity
* specialized color vision (cone-specific)
* contrast testing and night vision testing.

High-resolution spectral domain optical coherence tomography (SDOCT) images will be taken of the central retina using the Spectralis OCT unit. The values of visual function tested will be correlated with the findings on SDOCT (volume/amount of drusen present in early AMD).

There are no known risks to the subjects beyond what is normal for standard examinations of the eye, visual function testing and standard ocular photographic procedures.

DETAILED DESCRIPTION:
This prospective, exploratory study will be performed in multiple arms:

A. Arm 1: a pilot study of up to 40 patients (30 patients with dry age-related macular degeneration and 10 normal age-matched controls) in order to test 1) the feasibility of performing the visual function tests in this population and 2) test/retest reliability over 1-2 months. If the pilot study reveals that the visual function tests proposed are feasible and have high reliability, the larger study (Phase 2) will be subsequently performed.

B. Arm 2: a study of up to 160 patients (130 dry AMD patients and 32 controls) with the goal of evaluating the changes in visual function in dry AMD as compared to age-matched control subjects. Study will include patients determined on examination have dry AMD as well as age-matched normal control subjects without dry AMD. If two eyes satisfy the inclusion criteria, both eyes will be tested.

After consent is obtained following full explanation of the research, subjects will undergo the following non-invasive visual function testing: dark adaptation microperimetry with eye tracking, specialized color vision (cone specific), contrast testing and night vision testing. During the standard retina examination, color fundus photos will be taken using a Zeiss camera. Fundus Autoflorescence (FA), macular pigment optical density (MPOD) based on blue- green dual wave lenght FAF and high resolution spectral domain OCT(SDOCT) images will be taken of the central retina using the Heidelberg Spectralis OCT unit. The values of visula function tested will be correlated with the findings on SDOCT (volume/amount of drusen present in dry AMD).

During a testing day, the first patients first will undergo microperimetry testing, which incorporates an eye tracker that operates independently of the microperimeter and is able to compare results with a reference database of normal subjects. A Line Scanning Laser Ophthalmoscope (SLO) is used to capture confocal images of the retina. Using the SLO image, the operator can see the area to test. For follow-up examinations, the same area will be tested and the machine generates a report on change from previous examination. The test takes approximately 5 minutes.

Patients will then undergo cone specific vision testing. The cone contrast test (CCT) is a computer-based color test that rapidly identifies type (red, green, or blue) and severity (mild, moderate, and severe) of color deficiency, quantifies color performance, and allows early detection of acquired color deficiency. The automated test takes approximately 5 minutes to complete for all three cone tones; studies have shown impairment in blue and green cones in AMD. The system also provides tests for low contrast sensitivity night vision (simulate low lighting conditions, with darker background).

Using computerized visual acuity charts, the patients will also be tested for day and night glare and luminance. Using a dark adaptometer, the dark adaptation time will be measured. Subjects will also complete a quality of life questionnaire (NEI VFQ) and a low luminance questionnaire. The duration of each test can vary but typically lasts for 10-30 minutes.

A tube of blood about 5 ml will be collected from about 160 willing participants anytime during their study enrollment. The collected blood sample will be used for genetics studies associated with AMD. The samples will be stored here at the Duke Eye Center until all needed samples are obtained. All samples will be sent to Hoffman La Roche AG PDGE Functional Excellence, Biosample and Repository Management Evaluation of visual function impairments in patients with early dry age-related macular degeneration Basel, Switzerland for genetic testing.

Follow-up visual function testing will be performed at different time points depending on the Arm of the study: at 1-2 months for Arm 1 and approximately 6, 12, 18 and 24 months for Arm 2 using the same protocol, based on standard of care clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Capable and willing to provide consent
2. Has been diagnosed with dry age-related macular degeneration stages 1-3
3. At least 50 years of age

Exclusion Criteria:

1. Unable or unwilling to give consent
2. Under 50 years of age
3. Presence of retinal pathology such as central geographic atrophy, hemorrhage or retinal fluid, and other macular pathology other than AMD
4. Presence of dense cataracts in the study eye(s) that can affect visual function tests
5. Presence of glaucoma requiring treatment during the study and/or visual field defects
6. Presence retinal laser or surgical theraphy in study eye (s)
7. Any of other ocular condition requiring long-term theraphy or surgery during the study
8. Participant has photographically significant corneal or media opacities in either eye that would preclude adequate ophthalmic imaging and functional testing
9. Diagnosis of nystagmus that will interfere with testing
10. High myopia -8 Diopters or more severe
11. Participant has, in the opinion of the Investigator, any physical or mental condition that would increase the risk of participation in the stduy or may interfere with the study procedures, evaluations and outcome assessments.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified from patients of the Duke Eye Center presenting for ophthalmologic consultation. Patients with dry AMD are routinely available from this clinic and will be the primary study group.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2013-03; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in low luminance visual acuity | Arm 1: 1-2 months. Arm 2: 6, 12, 18 and 24 months

SECONDARY OUTCOMES:
Change in cone specific contrast sensitivity | Arm 1: 1-2 months. Arm 2: 6, 12, 18 and 24 months
Change in contrast sensitivity | Arm 1: 1-2 months. Arm 2: 6, 12, 18 and 24 months
Change in macular sensitivity on microperimetry | Arm 1: 1-2 months. Arm 2: 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Lad, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Cocce KJ, Stinnett SS, Luhmann UFO, Vajzovic L, Horne A, Schuman SG, Toth CA, Cousins SW, Lad EM. Visual Function Metrics in Early and Intermediate Dry Age-related Macular Degeneration for Use as Clinical Trial Endpoints. Am J Ophthalmol. 2018 May;189:127-138. doi: 10.1016/j.ajo.2018.02.012. Epub 2018 Mar 15. PMID 29477964
- [Result] Thompson AC, Luhmann UFO, Stinnett SS, Vajzovic L, Horne A, Toth CA, Cousins SW, Lad EM. Association of Low Luminance Questionnaire With Objective Functional Measures in Early and Intermediate Age-Related Macular Degeneration. Invest Ophthalmol Vis Sci. 2018 Jan 1;59(1):289-297. doi: 10.1167/iovs.17-22528. PMID 29340643